CLINICAL TRIAL: NCT05670353
Title: Cannabidiol in the Treatment of Women With Chronic Pelvic Pain Secondary to Endometriosis
Brief Title: Cannabidiol for the Treatment of Pelvic Pain in Endometriosis (DREAMLAND)
Acronym: DREAMLAND
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study was prematurely terminated due to the results of the interim analysis conducted, as outlined in the initial project plan.
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Omero Benedicto Poli Neto, Prof. Dr., University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021/10765-0
Record Dates: First submitted 2022-12-12; First posted 2023-01-04 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Endometriosis; Pelvic Pain
Keywords: Cannabis; Endometriosis; Pelvic Pain
MeSH Terms: conditions — Endometriosis; Pelvic Pain; Marijuana Abuse | interventions — Contraceptive Agents, Hormonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Volunteers, administrative staff, laboratory technicians, doctors who will carry out the assessments, and statisticians will be blind to the treatment group and will not know about the group treatment information.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabis Derivatives (Experimental): Cannabis Derivatives (98% CBD, 2% THC) will be given orally starting at 10 mg daily and up-titrated to a maximum dose of 150 mg daily. Dose up-titration will be based on clinical response or side effects, whichever comes first. After 63 days of treatment, gradual withdrawal will be performed during one week.
  All patients will take hormonal contraceptives, preferably progestagen-only.
  All participants will perform invasive and non-invasive procedures with the nursing team. The invasive will be blood collections, to evaluate laboratory parameters. The non-invasive ones refer to the measurement of height, weight, body temperature, and sleep pattern, as will pain threshold. In addition, they will be monitored through weekly self-assessment scales, applied remotely, electronically (cell phones or computers), with an estimated duration of ten minutes each, which will have their responses recorded in an electronic database, by the study coordination team.
  Interventions: Drug: Cannabis Derivatives; Drug: Hormonal Contraceptive Agents
- Placebo (Placebo Comparator): Placebo will be given at the same protocol described before. The bottle, label, color and density of the contents will be the same.
  All patients will take hormonal contraceptives, preferably progestagen-only. Then, at 70 days, there will be an open-label extension wherein all participants from control group will be offered a course of active treatment according to the same previous protocol.
  All participants will perform invasive and non-invasive procedures with the nursing team. The invasive will be blood collections, to evaluate laboratory parameters. The non-invasive ones refer to the measurement of height, weight, body temperature, and sleep pattern, as will pain threshold. In addition, they will be monitored through weekly self-assessment scales, applied remotely, electronically (cell phones or computers), with an estimated duration of ten minutes each, which will have their responses recorded in an electronic database, by the study coordination team.
  Interventions: Drug: Placebo; Drug: Hormonal Contraceptive Agents

INTERVENTIONS:
Drug: Cannabis Derivatives — CBD 10 mg (up-titrated until 150mg or adverse effects) daily for 9 weeks
  Arms: Cannabis Derivatives
Drug: Placebo — Placebo 10 mg (up-titrated until 150mg or adverse effects) daily for 9 weeks
  Arms: Placebo
Drug: Hormonal Contraceptive Agents — All participants will be given hormonal contraceptive.

SUMMARY:
The objective of this work is to conduct a randomized, double-blind, placebo-controlled clinical trial to assess the efficacy and safety of cannabis extract in women with endometriosis who have already undergone hormonal contraceptive treatment and surgery without satisfactory response.

DETAILED DESCRIPTION:
The Dreamland study is a two-arm, parallel-group, individually randomized (1:1 allocation ratio), controlled by disease stage, participant and investigator blinded, single-site superiority trial of oral cannabis extract (CBD). CBD will be given orally starting at 10 mg daily and up-titrated to a maximum dose of 150 mg daily. Dose up-titration will be based on clinical response or side effects, whichever comes first. After 63 days of treatment, gradual withdrawal will be performed during one week. Then, at 70 days, there will be an open-label extension wherein all participants from control group will be offered a course of CBD according to the same previous protocol.

This research intends to :

1. Assess whether the daily use of CBD, for nine weeks, will reduce the pain level of these women.
2. Assess whether the daily use of CBD, for nine weeks, will modify pain threshold.
3. Assess whether the daily use of CBD, for nine weeks, will interfere in psychological symptoms.
4. Assess the possible adverse effects of using CBD

ELIGIBILITY:
Inclusion Criteria:

* Women with chronic pelvic pain secondary to endometriosis surgically treated, with refractory symptoms, and who are taking complementary hormone therapy;
* Women over 18 years of age who wish to participate in the clinical trial;
* Willingness to voluntarily participate in the study to accept randomization to either of the two treatment arms;
* Participating exclusively in this clinical trial during the study period;
* Possess a telephone (cell or landline) that may be available to receive daily calls throughout the study period;
* Signature of the Free and Informed Consent Term (TCLE) approved by the Local Research Ethics Committee.

Exclusion Criteria:

* Chronic, severe or uncompensated medical conditions, such as: insulin-dependent diabetes (types 1 or 2); uncontrolled high blood pressure, lung disease such as asthma or other chronic obstructive pulmonary disease; hematological diseases, liver diseases, chronic kidney disease in advanced stage (grade 3, 4 and 5), metabolic disturbances and immunosuppression;
* Use of any medication with potential interaction with CBD/THC (such as chloroquine, clobazan, warfarin, or valproic acid) or history of undesirable reactions prior to the use of this medications;
* Inability to use oral medication;
* Pregnancy or lactation;
* History of alcohol or drug addiction;
* Smoking in the last three years;
* Marijuana use in the past three months or a lifetime history of dependence;
* Inability to cooperate with investigators due to cognitive impairment or mental status.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-01-03 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with pain change of 30% | Time points for assess: Week 1, Week 3, Week 4, Week 5, Week 7, Week 8, Week 9; Data will be reported through study completion, an average of 1 year
  Proportion of women with at least 30% of change in pain intensity. Pain intensity measured through visual analogue scale.
Proportion of patients with pain change of 50% | Time points for assess: Week 1, Week 3, Week 4, Week 5, Week 7, Week 8, Week 9; Data will be reported through study completion, an average of 1 year
  Proportion of women with at least 50% of change in pain intensity. Pain intensity measured through visual analogue scale.
Quantitative change in pain intensity | Time points for assess: Week 1, Week 3, Week 4, Week 5, Week 7, Week 8, Week 9; Data will be reported through study completion, an average of 1 year
  Absolute variation of pain intensity measured through visual analogue scale

SECONDARY OUTCOMES:
Pain threshold change | Day 0, Day 63
  Changes in the thermal peripheral pain thresholds: the range of temperatures at which a participant begins to perceive heat as painful: comparison between the beginning (day 0) and the end of the protocol (day 63).
Central sensitization change | Day 0, Day 63
  Changes in the score from Central Sensitization Inventory between the beginning (day 0) and the end of the protocol (day 63). Total scores ranging from 0-100. Higher scores mean a worse outcome. Score higher than 40 suggest central sensitization.
Brief measure for assessing generalized anxiety disorder | Day 0, Day 63
  Changes in the score from Generalized Anxiety Disorder (GAD7) scale between the beginning (day 0) and the end of the protocol (day 63). Total scores ranging from 0-21. Higher scores mean a worse outcome. Scores higher than 10 suggest generalized anxiety disorder.
Measure of the degree of depression severity | Day 0, Day 63
  Changes of scores for depressive symptoms over time during the study period (day 0-63) using Patient ́s Health Questionnaire-9 (PHQ-9). Total scores ranging from 0-27. Higher scores mean a worse outcome. Scores less than or equal to 4 suggest minimal depression.
Alanine aminotransferase (ALT) | Week 0, Week 1, Week 5, Week 9.
  Change in ALT concentration in plasma
Aspartate aminotransferase (AST) | Week 0, Week 1, Week 5, Week 9.
  Change in AST concentration in plasma
Glucose | Week 0, Week 1, Week 5, Week 9.
  Change in glucose concentration (glycemia) in plasma
Bilirubin | Week 0, Week 1, Week 5, Week 9.
  Change in bilirubin concentration in plasma
Cannabidiol (CBD) | Week 0, Week 1, Week 5, Week 9.
  Change in CBD concentration in plasma
Tetrahydrocannabinol (THC) | Week 0, Week 1, Week 5, Week 9.
  Change in THC concentration in plasma
Side effects | Week 0, Week 1 (Day 1, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7), Week 2, Week 3, Week 4, Week 5, Week 6, Week 7, Week 8, Week 9. Participants will be able to establish contact with a team doctor especially to report side effects.
  Occurrence of side effects over time during the study period (day 0-63)

CONTACTS AND LOCATIONS:
Locations (1):
- Center of Chronic Pelvic Pain and Gynecologic Endoscopy of Ribeirao Preto Medical School, University of Sao Paulo, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Immediately the following publication. No end date
Access Criteria: Researchers who provide a methodologically sound proposal. Depending on the level of the proposed use of data, approval by an independent review committee will be required for the identified purpose.